CLINICAL TRIAL: NCT07369128
Title: A Randomized, Dose-Ranging Trial of Propofol-Only and Dexmedetomidine-Propofol in Children Undergoing Magnetic Resonance Imaging
Brief Title: Propofol-Only Versus Dexmedetomidine-Propofol in Children Undergoing Magnetic Resonance Imaging
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Joseph Cravero, MD, Anesthesia, Critical Care and Pain Medicine, Principal Investigator, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IRB-P00052391
Record Dates: First submitted 2026-01-24; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: MRI Sedation; Pediatric Sedation; Propofol Dosage; Emergence Delirium, Anesthesia; Recovery Time; Dexmedetomidine
Keywords: pediatrics; sedation; dexmedetomidine; propofol; MRI
MeSH Terms: conditions — Emergence Delirium | interventions — Dexmedetomidine; Propofol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Propofol Only (P) (Active Comparator): If randomized to the P arm, the patient will receive a 2-4 mg/kg titrated IV bolus of propofol until sleep is induced. 250 mcg/kg/min infusion of IV propofol will then be started.
  Interventions: Drug: Propofol (IV) 2-4 mg/kg; Drug: Propofol (IV) Infusion 250 mcg/kg/min
- Dexmedetomidine (high)-Propofol (DHP) (Active Comparator): If randomized to the DHP arm, patient will receive an IV bolus of 1 mcg/kg of dexmedetomidine followed by a 1-2 mg/kg titrated IV bolus of propofol until sleep. 150 mcg/kg/min infusion of IV propofol will then be started. If not sedated within 10 minutes: 1-2 mg/kg bolus of propofol. If not sedated within 2 more minutes: 1-2 mg/kg bolus of propofol and increase propofol infusion to 200 mcg/kg/min (Can be titrated up to a maximum of 300 mcg/kg/min). If not sedated after 5 more minutes, record a technique failure and continue sedation at anesthesiologist's discretion.
  Interventions: Drug: Dexmedetomidine (IV) 1 mcg/kg; Drug: Propofol (IV) 1-2 mg/kg; Drug: Propofol (IV) Infusion 150 mcg/kg/min
- Dexmedetomidine (low)-Propofol (DLP) (Active Comparator): If randomized to the DLP arm, patient will receive an IV bolus of 0.5 mcg/kg of dexmedetomidine followed by a 1-2 mg/kg titrated IV bolus of propofol until sleep. 150 mcg/kg/min infusion of IV propofol will then be started. If not sedated within 10 minutes: 1-2 mg/kg bolus of propofol. If not sedated within 2 more minutes: 1-2 mg/kg bolus of propofol and increase propofol infusion to 200 mcg/kg/min (Can be titrated up to a maximum of 300 mcg/kg/min). If not sedated after 5 more minutes, record a technique failure and continue sedation at anesthesiologist's discretion.
  Interventions: Drug: Dexmedetomidine (IV) 0.5 mcg/kg; Drug: Propofol (IV) 1-2 mg/kg; Drug: Propofol (IV) Infusion 150 mcg/kg/min

INTERVENTIONS:
Drug: Dexmedetomidine (IV) 0.5 mcg/kg — If patient is randomized to the DLP arm, patient will receive an IV bolus of 0.5 mcg/kg dexmedetomidine over 5 minutes.
  Other Names: Precedex
  Arms: Dexmedetomidine (low)-Propofol (DLP)
Drug: Propofol (IV) 2-4 mg/kg — If patient is randomized to the P arm, patient will receive 2-4 mg/kg titrated, IV bolus of propofol until sleep is induced.
  Other Names: Diprivan
  Arms: Propofol Only (P)
Drug: Dexmedetomidine (IV) 1 mcg/kg — If patient is randomized to the DHP arm, patient will receive an IV bolus of 1 mcg/kg dexmedetomidine over 5 minutes.
  Other Names: Precedex
  Arms: Dexmedetomidine (high)-Propofol (DHP)
Drug: Propofol (IV) 1-2 mg/kg — If the patient is randomized to the DLP or DHP arm, following the dexmedetomidine bolus, the patient will receive a titrated, IV bolus of 1-2 mg/kg propofol.
  Other Names: Diprivan
  Arms: Dexmedetomidine (high)-Propofol (DHP); Dexmedetomidine (low)-Propofol (DLP)
Drug: Propofol (IV) Infusion 250 mcg/kg/min — If the patient is randomized to the P arm, following the bolus of propofol, the patient will be started on an IV propofol infusion of 250 mcg/kg/min.
  Other Names: Diprivan
  Arms: Propofol Only (P)
Drug: Propofol (IV) Infusion 150 mcg/kg/min — If the patient is randomized to the DLP or DHP arm, following the titrated propofol bolus, the patient will be started on an IV propofol infusion of 150 mcg/kg/min.
  Other Names: Diprivan
  Arms: Dexmedetomidine (high)-Propofol (DHP); Dexmedetomidine (low)-Propofol (DLP)

SUMMARY:
The most common imaging procedure requiring sedation/anesthesia for the pediatric population is magnetic resonance imaging (MRI). However, the optimal anesthetic/sedation plan has not been determined for these procedures. Historically, common medications have included the use of pentobarbital and propofol, but in 2015, publication in the New England Journal of Medicine highlighted the accumulating evidence for the possible neurotoxic effects of these types of anesthetics in animal models and a collection of epidemiologic studies in humans. Although these initial possibilities have since been proven as less of a concern, in the interim, data has shown that alternative sedative agents, such as dexmedetomidine, may not have the same neurotoxic effect and could possibly even provide neuroprotection. Dexmedetomidine also possesses other beneficial traits such as reducing risks of pulmonary atelectasis or upper airway collapse, typically found with the administration of propofol.

A concern raised by previous studies has been the possibility that the addition of dexmedetomidine could increase recovery times, leading to disruptions in workflow. Although it has been shown that large doses of dexmedetomidine exposure may lead to longer PACU stays, it is uncertain whether a small dose of dexmedetomidine would have such a significant impact. Based on the investigators' pilot trial6, the investigators found that a bolus of 1 mcg/kg dose of dexmedetomidine with a bolus of titrated propofol of 2-3 mg/kg and an infusion of propofol of 100 mcg/kg/min provided adequate sedation for successful scans, reduced propofol (infusion) exposure by 60%, and did not significantly increase recovery times.

Finally, there is a paucity in literature for studies examining a range of doses subsequently; often, a control group is compared to a single, self-selected dose of choice. Here, the investigators hope to provide a range of doses to minimize selection bias in our study design and determine the dose that would provide the optimal sedation for these scans and minimize excess anesthetic exposure.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting as outpatients, scheduled to receive an anesthetic for MRI of brain, body (spine, chest, abdomen, and/or pelvis) and/or extremity (arm and/or leg).
* Patients must be a candidate for the sedation technique described in this study with a natural airway. This decision will be made by a staff member of the Department of Anesthesiology.
* Between 1 and 12 years of age.
* ASA status I, II, or III

Exclusion Criteria:

* Inpatient at BCH
* Diagnosis of a difficult airway, severe obstructive sleep apnea that is not compatible with spontaneous ventilation in a supine position, or requires an oral airway.
* Congenital heart disease or history of dysrhythmia.
* Taking digoxin or beta-blocker
* Anxiolytic medication is ordered before the MRI (e.g., midazolam or ketamine).
* History or a family (parent or sibling) history of malignant hyperthermia.
* Allergy to or has a contraindication to propofol or dexmedetomidine.
* Tracheostomy or other mechanical airway device present
* Received within the past 12 hours an oral or intravenous alpha-adrenergic, beta-adrenergic agonist, or antagonist drugs (e.g., clonidine, propranolol, albuterol).
* Patient is not scheduled to receive anesthesia-sedation care or is noted to "try-without anesthesia" for the MRI
* Patient has significant developmental or psychological delays
* Patient scheduled for scan of duration <30 minutes or >90 minutes

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 105 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Total Propofol (mcg/kg/min) consumption | Up to 120 minutes or from induction of anesthesia/sedation to end of MRI scan
  The total amount of propofol (mcg/kg/min) consumed will be measured for the duration of anesthesia time for the P, DLP, and DHP arms.

SECONDARY OUTCOMES:
Peak Pediatric Anesthesia Emergence Delirium (PAED) Score | Up to 180 minutes or duration of PACU stay
  The peak (highest) PAED score will be obtained in the post-anesthesia recovery area (PACU).
Incidence of Adverse Events | Up to 240 minutes or from induction of anesthesia/sedation to immediately during recovery
  Arterial desaturation, airway obstruction, hypotension and bradycardia
Incidences of Patient Movements/MRI Interruptions | Up to 90 minutes or duration of MRI scan
  If patient moved during their MRI and caused an interruption of the scan.
Incidence of Technique Failure | Up to 120 minutes or from induction of anesthesia/sedation to end of MRI scan
  Lack of adequate sedation for MRI scan in spite of the sedation as described above (based on anesthesiologist's discretion or PSSS)
Case Duration | Up to 90 minutes or duration of MRI scan
  Total number of minutes in the MRI scanner
Post Anesthesia Care Unit (PACU) Duration | Up to 180 minutes or duration of PACU stay
  Total number of minutes in the PACU

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Cravero, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nagoshi M, Reddy S, Bell M, Cresencia A, Margolis R, Wetzel R, Ross P. Low-dose dexmedetomidine as an adjuvant to propofol infusion for children in MRI: A double-cohort study. Paediatr Anaesth. 2018 Jul;28(7):639-646. doi: 10.1111/pan.13400. Epub 2018 Jun 7. PMID 29882298
- [Background] Ramaprasannakumar SK, Bhadrinarayan V, Venkataramaiah S. The Effectiveness of Three Regimens of Sedation for Children Undergoing Magnetic Resonance Imaging: A Clinical Study. Anesth Essays Res. 2022 Jul-Sep;16(3):345-352. doi: 10.4103/aer.aer_45_22. Epub 2022 Dec 9. PMID 36620110
- [Background] Boriosi JP, Eickhoff JC, Klein KB, Hollman GA. A retrospective comparison of propofol alone to propofol in combination with dexmedetomidine for pediatric 3T MRI sedation. Paediatr Anaesth. 2017 Jan;27(1):52-59. doi: 10.1111/pan.13041. Epub 2016 Oct 25. PMID 27779360
- [Background] Vinson AE, Peyton J, Kordun A, Staffa SJ, Cravero J. Trends in Pediatric MRI sedation/anesthesia at a tertiary medical center over time. Paediatr Anaesth. 2021 Sep;31(9):953-961. doi: 10.1111/pan.14225. Epub 2021 Jun 22. PMID 34036674
- [Background] Kim SY, Booth JM, Staffa SJ, Kordun A, Yu J, Cravero JP. A dose-ranging pilot trial of dexmedetomidine-propofol in children undergoing magnetic resonance imaging. J Anesth. 2025 Dec;39(6):989-994. doi: 10.1007/s00540-025-03511-z. Epub 2025 May 11. PMID 40349256
- [Background] Rappaport BA, Suresh S, Hertz S, Evers AS, Orser BA. Anesthetic neurotoxicity--clinical implications of animal models. N Engl J Med. 2015 Feb 26;372(9):796-7. doi: 10.1056/NEJMp1414786. PMID 25714157
- [Background] Mallory MD, Travers C, Cravero JP, Kamat PP, Tsze D, Hertzog JH. Pediatric Sedation/Anesthesia for MRI: Results From the Pediatric Sedation Research Consortium. J Magn Reson Imaging. 2023 Apr;57(4):1106-1113. doi: 10.1002/jmri.28392. Epub 2022 Aug 12. PMID 36173243